CLINICAL TRIAL: NCT04752748
Title: Power Doppler in Hand Joints is a Predictor of Therapeutic Failure in Women With Early Rheumatoid Arthritis Naive for Treatment
Brief Title: Power Doppler in Hand Joints of Early RA Patients
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Karine Rodrigues da Luz, Principal Investigator, Federal University of São Paulo
Other Study IDs: 106108
Record Dates: First submitted 2021-02-10; First posted 2021-02-12 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Early Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Drug Therapy, Computer-Assisted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Woman with Early Rheumatoid Arthritis
  Interventions: Drug: Drug protocol

INTERVENTIONS:
Drug: Drug protocol — The following drug scheme was carried out: The patients began with methotrexate (MTX) 15 mg / week, which was increased to 25 mg / week until week 12. Subsequent steps for patients with an insufficient response (DAS28 score> 3.2 and the Physician's Global Assessment (PGA)> 4.0 [0-10 cm]) were leflunomide 20mg / day with MTX 15 mg / week from week 12 to week 24 and adalimumab twice a month and MTX 15mg / week from week 24 to week 48. The use of 5mg folic acid was advised once a week during the 48 weeks of the study. Three treatment failures were considered over these 48 weeks:
  * Failure 1: failure of the first DMARD (MTX) in week 12.
  * Failure 2: failure of the second DMARD (leflunomide) at week 24
  * Failure 3: failure of the first immunobiological (adalimumab) at week 48.

SUMMARY:
It is a prospective case-control study with women diagnosed early rheumatoid arthritis. Three therapeutic failures were considered: failure 1 - to the first Disease-modifying antirheumatic drugs (DMARDs) (methotrexate); failure 2 - to the second DMARDs (leflunomide) and failure 3 - to the first immunobiological drugs (adalimumab). Ultrasound was performed bilaterally on the 2nd and 3rd metacarpophalangeal joints (MCFs), proximal interphalangeal joints (IFPs), and wrists (US10). Ultrasound measurements (qualitative and semi-quantitative) evaluated: 1 - inflammatory: synovial and tenosynovial proliferation in gray scale and power Doppler (0-3); 2 - joint damage: bone erosion (qualitative and semi-quantitative) and cartilage damage (qualitative and semi-quantitative). Clinical and laboratory variables were also assessed blindly at baseline and after 12, 24 e 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* early rheumatoid arthritis fulfilment of the 2010 ACR/EULAR RA classification criteria;
* age between 18-65 years;
* female gender,
* naive for treatment.

Exclusion Criteria:

* use of oral > 10 mg/d glucocorticoid in the previous three weeks;
* serum aspartate aminotransferase or alanine aminotransferase level > 3 times the upper limit of normal;
* bone marrow, auto-imune, lymphoproliferative or infectious diseases;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman diagnosed eith early rheumatoid arthritis naive for treatment
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in Synovial blood flow (power doppler) | Baseline, after 4, 12, 24 and 48 weeks
  Measured in ultrasound examination

SECONDARY OUTCOMES:
Change in Synovial Proliferation | Baseline, after 4, 12, 24 and 48 weeks
  Measured in ultrasound examination
Changes in Tenosynovitis | Baseline, after 4, 12, 24 and 48 weeks
  Measured in ultrasound examination
Changes in Joint Damage | Baseline, after 4, 12, 24 and 48 weeks
  Measured in ultrasound examination
Changes in C-reactive protein level (mg/liter) | Baseline, after 4, 12, 24 and 48 weeks
  Measured in blood test
Changes in erythrocyte sedimentation rate level (mm/hour) | Baseline, after 4, 12, 24 and 48 weeks
  Measured in blood test
Changes in function | Baseline, after 4, 12, 24 and 48 weeks
  Measured by Health Assessment Questionnaire
Changes in upper limb function | Baseline, after 4, 12, 24 and 48 weeks
  Measured by Disabilities of the Arm, Shoulder and Hand Questionnaire
Changes in disease activity score | Baseline, after 4, 12, 24 and 48 weeks
  Measured by disease activity score 28

REFERENCES:
- [Derived] da Luz KR, Natour J, Pinheiro MM, Petterle GS, Dos Santos MF, Fernandes ADRC, Furtado RNV. Power Doppler in hand joints predicts therapeutic failure in treatment-naive women with early rheumatoid arthritis: A prospective study. Clinics (Sao Paulo). 2025 Mar 1;80:100593. doi: 10.1016/j.clinsp.2025.100593. eCollection 2025. PMID 40023888